CLINICAL TRIAL: NCT05828069
Title: Phase 2 Study of Tovorafenib (DAY101) in Relapsed and Refractory Langerhans Cell Histiocytosis
Brief Title: A Study With Tovorafenib (DAY101) as a Treatment Option for Progressive, Relapsed, or Refractory Langerhans Cell Histiocytosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-06282; NCI-2022-06282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANHL2121 (Other: Children's Oncology Group); ANHL2121 (Other: CTEP); U10CA180886 (NIH); NCT05287295 (obsolete NCT alias)
Record Dates: First submitted 2023-04-21; First posted 2023-04-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Langerhans Cell Histiocytosis; Refractory Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Specimen Handling; Biopsy; Spinal Puncture; tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tovorafenib) (Experimental): Patients receive tovorafenib PO QW on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MUGA or ECHO scans, and FDG-PET or CT throughout the trial, and collection of blood and urine samples on study. Patients with suspicion of bone marrow and/or central nervous system involvement will also undergo bone marrow biopsy and aspiration and lumbar puncture on study and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan; Procedure: Lumbar Puncture; Procedure: Multigated Acquisition Scan; Drug: Tovorafenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan — Undergo FDG-PET imaging
  Other Names: FDG PET/CT
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Tovorafenib — Given PO
  Other Names: BIIB 024; BIIB-024; BIIB024; DAY 101; DAY-101; DAY101; MLN 2480; MLN-2480; MLN2480; Ojemda; pan-RAF Kinase Inhibitor DAY101; TAK 580; TAK-580; TAK580

SUMMARY:
This phase II trial tests the safety, side effects, best dose and activity of tovorafenib (DAY101) in treating patients with Langerhans cell histiocytosis that is growing, spreading, or getting worse (progressive), has come back (relapsed) after previous treatment, or does not respond to therapy (refractory). Langerhans cell histiocytosis is a type of disease that occurs when the body makes too many immature Langerhans cells (a type of white blood cell). When these cells build up, they can form tumors in certain tissues and organs including bones, skin, lungs and pituitary gland and can damage them. This tumor is more common in children and young adults. DAY101 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Using DAY101 may be effective in treating patients with relapsed or refractory Langerhans cell histiocytosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine overall response rate (ORR) for children and young adults with relapsed or refractory BRAFV600E positive (cohort 1) and BRAFV600E negative (cohort 2) Langerhans cell histiocytosis (LCH) treated with tovorafenib (DAY101) after 2 cycles and must be maintained 4 weeks later.

SECONDARY OBJECTIVES:

I. To determine nature and severity of adverse events in patients treated with tovorafenib (DAY101) for relapsed or refractory LCH.

II. To describe event-free survival (EFS) at 1 year in children and young adults with relapsed and refractory LCH treated with tovorafenib (DAY 101) for up to 1 year.

III. To determine durability of response in children and young adults with relapsed or refractory LCH treated with tovorafenib (DAY101) following cessation of therapy in patients with complete response (CR) at 1 year.

IV. To describe progression-free (and relapse-free) survival (PFS) and overall survival (OS) in children and young adults with relapsed or refractory LCH treated with tovorafenib (DAY101) for up to 1 year.

EXPLORATORY OBJECTIVES:

I. To determine potential role of pathogenic tumor mutation in response to tovorafenib (DAY101), and to evaluate changes in bone marrow and peripheral blood cell populations carrying pathogenic mutations in response to tovorafenib (DAY101) therapy.

Ia. To define somatic mutations in LCH lesion biopsies; Ib. To determine impact of tovorafenib (DAY101) on bone marrow and blood BRAFV600E+ mononuclear cells; Ic. To determine impact of tovorafenib (DAY101) on cerebral spinal fluid and disease response; Id. To determine the performance of standardized immunohistochemical analysis of LCH lesion biopsies.

II. To compare performance of LCH-specific response criteria to Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

III. To describe the pharmacokinetics of tovorafenib (DAY101) when administered to pediatric and young adult patients with relapse or refractory LCH.

OUTLINE: This is a dose escalation study of tovorafenib followed by a phase II trial.

Patients receive tovorafenib orally (PO) once weekly (QW) on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo multi-gated acquisition (MUGA) or echocardiography (ECHO) scans, and fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) or computed tomography (CT) throughout the trial, and collection of blood and urine samples on study. Patients with suspicion of bone marrow and/or central nervous system involvement will also undergo bone marrow biopsy and aspiration and lumbar puncture on study and during follow up.

After completion of study treatment, patients are followed up at 28 days, months 3, 6, 9, and 12, and then at 2 years post cycle 12.

ELIGIBILITY:
Inclusion Criteria:

* 180 days- < 22 years (at time of study enrollment)
* Patient must have a body surface area of ≥ 0.3 m^2
* Patients with progressive, relapsed, or recurrent LCH with measurable disease at study entry

  * Patients must have had histologic verification of LCH (from either original diagnosis or relapse/progression) at the time of study entry

    * Tissue confirmation of relapse is recommended but not required.
    * Pathology report must be submitted for central confirmation of diagnosis within 7 days of enrollment.
    * Formalin-fixed paraffin-embedded (FFPE) blocks or unstained slides (initial diagnosis and/or subsequent biopsies) will be required for retrospective central confirmation of diagnosis and molecular studies
    * Patients with mixed histiocytic disorders (e.g. LCH with juvenile xanthogranuloma) may be included
  * Patients must have measurable disease
  * Patients must have progressive or refractory disease or experience relapse after at least one previous systemic treatment strategy
  * Pathogenic somatic mutation detected in genes encoding tyrosine kinase receptors (CSFR1, ERBB3 or ALK), RAS or RAF (may be from original or subsequent biopsy or peripheral blood/bone marrow aspirate). Clinical mutation reports may include quantitative polymerase chain reaction (PCR) (e.g. BRAFV600E) and/or Sanger or next generation sequencing. Immunohistochemistry (e.g. VE1 antibody for BRAFV600E) alone is not sufficient
* Participant must be able to take an enteral dose and formulation of medication. Study medication is only available as an oral suspension or tablet, which may be taken by mouth or other enteral route such as nasogastric, jejunostomy, or gastric tube
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50% for patients =< 16 years of age
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Myelosuppressive chemotherapy: Patients must not have received within 14 days of entry onto this study
* Investigational agent or any other anticancer therapy not defined above: Patients must not have received any investigational agent or any other anticancer therapy (including MAPK pathway inhibitor) for at least 14 days prior to planned start of tovorafenib (DAY101)
* Radiation therapy (RT): Patient must not have received RT within 2 weeks after the last dose fraction of RT
* Patients must have fully recovered from any prior surgery
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, targeted inhibitor, and/or radiotherapy with toxicities reduced to grade 1 or less (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0)
* Steroids: =< 0.5 mg/kg/day of prednisone equivalent (maximum 20 mg/day) averaged during the month prior to study enrollment is permissible
* Strong inducers or inhibitors of CYP2C8 are prohibited for 14 days before the first dose of tovorafenib (DAY101) and from planned administration for the duration of study participation
* Medications that are breast cancer resistant protein (BCRP) substrates that have a narrow therapeutic index are prohibited for 14 days before the first dose of tovorafenib (DAY101) and for the duration of study participation
* Peripheral absolute neutrophil count (ANC) >= 750/uL unless secondary to bone marrow involvement, in such cases bone marrow involvement must be documented (must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* Platelet count >= 75,000/uL (unsupported/without transfusion within the past 7 days) (must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* Patients with marrow disease must have platelet count of >= 75,000/uL (transfusion support allowed) and must not be refractory to platelet transfusions. Bone marrow involvement must be documented
* Hemoglobin >= 8 g/dL (unsupported/without transfusion within the past 7 days). Patients with marrow disease must have hemoglobin >= 8 g/dL (transfusion support allowed). Bone marrow involvement must be documented
* Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g., Neulasta [registered trademark]) or 7 days for short-acting growth factor
* A serum creatinine based on age/sex as follows (must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)

  * Age: 6 months to < 1 year; Maximum Serum Creatinine (mg/dL):= 0.5 mg/dl (male and female)
  * Age: 1 to < 2 years; Maximum Serum Creatinine (mg/dL): = 0.6 mg/dl (male and female)
  * Age: 2 to < 6 years; Maximum Serum Creatinine (mg/dL): = 0.8 mg/dl (male and female)
  * Age: 6 to < 10 years; Maximum Serum Creatinine (mg/dL): = 1.0 mg/dl (male and female)
  * Age: 10 to < 13 years; Maximum Serum Creatinine (mg/dL): = 1.2 mg/dl (male and female)
  * Age: 13 to < 16 years; Maximum Serum Creatinine (mg/dL): = 1.5 mg/dl (male) and 1.4 mg/dl (female)
  * Age: >= 16 years; Maximum Serum Creatinine (mg/dL): = 1.7 mg/dl (male) and 1.4 mg/dl (female)
  * OR- a 24 hour urine creatinine clearance >= 50 mL/min/1.73 m^2
  * OR- a glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* Alanine aminotransferase (ALT) =< 3 x ULN for age (must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* Serum albumin >= 2 g/dl must be performed within 7 days prior to enrollment, must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* For patients with liver disease caused by their histiocytic disorder (as evaluated on radiographic imaging or biopsy): patients may be enrolled with abnormal bilirubin, aspartate aminotransferase (AST), ALT and albumin with documentation of histiocytic liver disease
* Fractional shortening (FS) of >= 25% or ejection fraction of >= 50%, as determined by echocardiography or multigated acquisition scan (MUGA) within 28 days prior to study enrollment. Depending on institutional standard, either FS or left ventricular ejection fraction (LVEF) is adequate for enrollment if only one value is measured; if both values are measured, then both values must meet criteria above (must be obtained within 28 days prior to enrollment and start of protocol therapy) (repeat if necessary)
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination; unless it is due to underlying pulmonary LCH
* Central Nervous System Function Defined As:

  * Patients with seizure disorder may be enrolled if well controlled
  * Central nervous system (CNS) toxicity =< Grade 2
* Human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial unless antiretroviral therapy interacts with the metabolism of tovorafenib (DAY101) and cannot safely be changed to antivirals that do not interact with study medication
* All patients and/or their parent(s) or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* LCH arising along with other hematologic malignancy (e.g. mixed LCH with acute lymphoblastic leukemia) or any history of non-histiocytic malignancy
* Disease scenarios as below will be excluded

  * Skin-limited disease
  * Gastrointestinal (GI) tract involvement only (those that have disease that can be determined by endoscopic biopsies only)
  * LCH-associated neurodegeneration (LCH-ND) without parenchymal lesions or other systemic lesions
* Patients with activating mutations in MAP2K1 are not eligible for this study due to drug target specificity. Mutation status will be submitted to study team within 7 days of enrollment
* Refractory nausea and vomiting, malabsorption, or external biliary shunt that would preclude adequate absorption of tovorafenib (DAY101)
* Uncontrolled systemic bacterial, viral, or fungal infection
* Major surgical procedure or significant traumatic injury within 14 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study. Placement of a vascular access device or minor surgery is permitted within fourteen (14) days of study enrollment (provided that the wound has healed)
* History of significant bowel resection that would preclude adequate absorption or other significant malabsorptive disease
* Ophthalmologic considerations: Patients with known significant ophthalmologic conditions or known risk factors for retinal vein occlusion (RVO) or central serous retinopathy (CSR) are not eligible
* History of solid organ or hematopoietic bone marrow transplantation
* Clinically significant active cardiovascular disease, or history of myocardial infarction, or deep vein thrombosis/pulmonary embolism within 6 months prior to enrollment, ongoing cardiomyopathy, or current prolonged QT interval > 440 ms based on triplicate electrocardiogram (ECG) average
* History of Grade >= 2 CNS hemorrhage or history of any CNS hemorrhage within 28 days of study entry
* History of any drug reaction with eosinophilia and systemic symptoms (DRESS) syndrome or Stevens Johnsons syndrome (SJS) or who are allergic to tovorafenib (DAY101) or any of its components
* CTCAE version (V.) 5.0 Grade 3 symptomatic creatinine kinase (CPK) elevation (> 5 x ULN)
* Female patients who are pregnant are ineligible. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants are ineligible
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation are ineligible. Women of childbearing potential must use non-hormonal contraception during tovorafenib treatment and for at least 28 days after the last dose. Men should use effective contraception and must not father a child while taking tovorafenib and for 14 days after the last dose

Ages: 180 Days to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicity (dose finding phase) | Up to 28 days
  Will be analyzed descriptively.
Overall response rate (phase II) | After 2 cycles of therapy (each cycle is 28 days)
  Will be assessed using minimax Simon's two-stage designs in each of the BRAFV600E and non-BRAFV600E cohorts separately. The two arms will not be directly compared. The 95% confidence interval for the overall response rate will be adjusted for the two-stage design.

SECONDARY OUTCOMES:
Event free survival rate | At 1 and 2 years
  Will be estimated by the Kaplan-Meier method beginning at study enrollment. Will be evaluated two years after enrollment of the last patient on the trial and estimates at specific timepoints will be presented along with log-log transformed 95% confidence intervals. Events are defined as relapse/progression, second malignant neoplasm, or death.
Progression free survival rate | Up to 2 years
  Will be estimated by the Kaplan-Meier method beginning at study enrollment. Will be evaluated by two years after enrollment of the last patient on the trial and estimates at specific timepoints will be presented along with log-log transformed 95% confidence intervals.
Duration of response rate | After 12 months of therapy. From the scan confirming the complete response or partial response (whichever is recorded first), until the first occurrence of recurrent or progressive disease or death (event) or last known status on trial
  Response is based on modified Response Evaluation Criteria for Solid Tumors (RECIST)/Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) consistent with other recent pediatric Langerhans Cell Histiocytosis trials (NCT02670707 and NCT04079179) and adult histiocytosis trials with MAPK inhibitors. Comparison of response assessed via RECIST versus (vs.) PERCIST will be analyzed by displaying two-way tables of the responses with no formal statistical testing.
Overall survival rate | Up to 2 years
  Will be estimated by the Kaplan-Meier method beginning at study enrollment. Will be evaluated two years after enrollment of the last patient on the trial and estimates at specific timepoints will be presented along with log-log transformed 95% confidence intervals.

OTHER OUTCOMES:
Percent peripheral blood mononuclear cells with mutated allele | Up to 2 years
  Will be analyzed descriptively using logistic regression with complete response/progressive response vs. stable disease/progressive disease as the response variable.

CONTACTS AND LOCATIONS:
Overall Officials: Carl E Allen, Principal Investigator — Children's Oncology Group
Locations (113):
- United States (100):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm